CLINICAL TRIAL: NCT02962440
Title: A Single Centre, Open Label Trial Investigating the Absorption, Metabolism and Excretion of Somapacitan After Single Subcutaneous Dosing in Healthy Male Subjects
Brief Title: A Trial Investigating the Absorption, Metabolism and Excretion of Somapacitan After Single Dosing in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NN8640-4237; 2016-000096-24 (EudraCT Number); U1111-1178-1251 (Other: World Health Organization (WHO))
Record Dates: First submitted 2016-11-09; First posted 2016-11-11 (Estimated); Last update posted 2017-06-07 (Actual); Status verified 2017-06

CONDITIONS: Healthy
MeSH Terms: interventions — somapacitan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Somapacitan (Experimental)
  Interventions: Drug: somapacitan

INTERVENTIONS:
Drug: somapacitan — All subjects will receive one subcutaneous (s.c., under the skin) dose of somapacitan containing [3H]-somapacitan

SUMMARY:
This trial is conducted in Europe. The aim of the trial is to investigate the absorption, metabolism and excretion of somapacitan after single subcutaneous dosing in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male, aged 45-64 years (both inclusive) at the time of signing informed consent
* Body mass index (BMI) 20.0-29.9 kg/m^2 (both inclusive)
* Considered to be generally healthy based on the medical history, physical examination, and the results of vital signs, electrocardiogram and clinical laboratory tests performed during the screening visit, as judged by the investigator

Exclusion Criteria:

* Male of reproductive age who or whose partner(s) is not willing to use adequate contraceptive methods (adequate contraceptive measures as required by local regulation or practice) for at least 4 months after dosing or male who is not willing to refrain from donating semen for at least 4 months after dosing. Acceptable forms of prevention include complete sexual abstinence, surgically sterilisation, that the subject uses a condom during intercourse or that the partner practices adequate contraception (risk of pregnancy must be lower than 1%).
* Use of prescription or non-prescription products, including herbal products and non-routine vitamins, within 14 days prior to screening. Occasional use of paracetamol is permitted.
* Any blood draw in excess of 25 mL in the past 30 days, or donation of blood or plasma in excess of 400 mL within the 90 days preceding screening.

Ages: 45 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2016-11; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Total amount of [3H]-somapacitan related material excreted in urine (% of dose) | Assessed up to 35 days after trial product administration
Total amount of [3H]-somapacitan related material excreted in faeces (% of dose) | Assessed up to 35 days after trial product administration
Total amount of [3H]-somapacitan related material excreted in expired air (% of dose) | Assessed up to 35 days after trial product administration

SECONDARY OUTCOMES:
Total recovery of administered 3H label (sum of urine, faeces and expired air) | Assessed up to 36 days after trial product administration
Blood to plasma ratio of [3H]-somapacitan related material | Assessed up to 36 days after trial product administration

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Groningen, Netherlands

REFERENCES:
- [Derived] Helleberg H, Bjelke M, Damholt BB, Pedersen PJ, Rasmussen MH. Absorption, metabolism and excretion of once-weekly somapacitan, a long-acting growth hormone derivative, after single subcutaneous dosing in human subjects. Eur J Pharm Sci. 2021 Dec 1;167:106030. doi: 10.1016/j.ejps.2021.106030. Epub 2021 Oct 1. PMID 34601071